CLINICAL TRIAL: NCT00506779
Title: A Phase I/II Study of Gleevec/Taxol in Patients With Newly Diagnosed Stage IIIC or IV or Recurrent (Any Stage) Uterine Papillary Serous Carcinoma (UPSC)
Brief Title: Gleevec/Taxol for Patients With Uterine Papillary Serous Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the study was terminated early due to poor enrollment
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GYN03-0177; NCI-2012-01549 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Uterine Cancer
Keywords: Uterine Papillary Serous Carcinoma; Uterine Cancer; UPSC; Taxol; Paclitaxel; Gleevec; Imatinib Mesylate; STI571
MeSH Terms: conditions — Uterine Neoplasms | interventions — Imatinib Mesylate; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I: Paclitaxel + Imatinib Mesylate (Experimental): Phase I MTD using oral dose Imatinib Mesylate escalation 400, 500, 600 mg daily; Paclitaxel 175 mg/m^2 every 21 days
  Interventions: Drug: Imatinib Mesylate; Drug: Paclitaxel
- Phase II: Paclitaxel Alone or Pacliataxel + Imatinib Mesylate (Experimental): Intended randomization of Paclitaxel alone or Paclitaxel + Imatinib Mesylate; the study was terminated early due to poor enrollment and all patients are no longer being treated or followed. Single treatment arm MTD using oral dose Imatinib Mesylate escalation = 500 mg daily; Paclitaxel 175 mg/m^2 every 21 days
  Phase II, (Arm 1) = Paclitaxel 175 mg/m^2 every 21 days Phase II, (Arm 2) Paclitaxel 175 mg/m^2 every 21 days+ Imatinib Mesylate MTD using oral dose Imatinib Mesylate escalation = 500 mg daily
  Interventions: Drug: Imatinib Mesylate; Drug: Paclitaxel

INTERVENTIONS:
Drug: Imatinib Mesylate — Phase I = Maximum tolerated dose (MTD) derived from dose escalation of 400, 500, 600 mg by mouth daily
  Other Names: Gleevec; STI571; Imatinib; NSC-716051
Drug: Paclitaxel — 175 mg/m^2 by vein over 3 Hours every 21 Days
  Other Names: Taxol

SUMMARY:
Objectives:

* To determine the maximum tolerated dose (MTD) of imatinib mesylate in combination with fixed dose paclitaxel in patients with stage IIIC, IV or recurrent uterine papillary serous carcinoma.
* To determine the nature and degree of toxicity of imatinib mesylate and paclitaxel in this cohort of patients.
* To determine the efficacy of imatinib mesylate and paclitaxel in patients with stage IIIC, IV or recurrent uterine papillary serous carcinoma whose tumor expresses either c-Kit, PDGFR or abl.

DETAILED DESCRIPTION:
Before possible study participants can receive treatment with imatinib mesylate and paclitaxel, their tumor tissue that was previously collected (at the surgery to diagnose your tumor) will be tested for the following three biomarkers: c-Kit, PDGFR-B, and Abl. Those participants who have at least one positive biomarker will be eligible for treatment on this study.

Paclitaxel is a chemotherapy drug used in the treatment of ovarian cancer. Imatinib mesylate is a medication that blocks several proteins that are important in the development of cancer.

Before treatment starts, you will have a complete physical exam, routine blood tests (about 2-3 teaspoons), an electrocardiogram (ECG--a test to measure the electrical activity of the heart). You will have an echocardiogram (an ultrasound test used to visualize the structures of the heart), a chest x-ray, and a CT scan or MRI of the abdomen and pelvis. Women who are able to have children must have a negative blood pregnancy test.

Routine blood tests (about 2 teaspoons) will be done weekly during treatment, and before each course of therapy, which is every 3 weeks. A complete checkup including evaluation of side effects, will also be done before each course of therapy and at the end of therapy (3 weeks after treatment ends).

There are two phases to this study, Phase I and Phase II. If you are assigned to Phase 1, you will receive treatment with imatinib mesylate and paclitaxel. Phase 1 will study 3 different doses of imatinib mesylate in combination with a fixed dose of paclitaxel. The Phase I part of the study will help researchers learn the most effective dose of imatinib mesylate to be used in combination with paclitaxel. All participants in Phase 1 will receive one of three doses of imatinib mesylate to be given with a standard dose of paclitaxel. You will be assigned to a specific dose level based on the number of participants treated at the time of your enrollment.

The Phase II portion of the study will begin only after the most effective dose of imatinib mesylate has been determined.

If you are assigned to Phase II, you will be randomly assigned (as in the toss of a coin) to one of two treatment groups. Participants in one group will receive treatment with paclitaxel only (every 21 days). Participants in the second group will receive treatment with paclitaxel (every 21 days) along with imatinib mesylate (every day). The dose level of imatinib mesylate that you receive will be the same as the dose used during Phase I. The computer-generated assignment will favor the treatment group which is more effective. For example, if the combination of paclitaxel and imatinib mesylate is more effective than paclitaxel alone, then more patients will be selected to receive the combination therapy.

You will receive paclitaxel by vein over 3 hours every 21 days. Those participants who are assigned treatment with both paclitaxel and imatinib mesylate will begin taking imatinib mesylate the day after the first dose of paclitaxel. A single dose of imatinib mesylate will be taken by mouth every day.

Evaluation of tumor response (for participants who already have the disease) will be determined by CT scan or MRI and chest x-ray (patients with chest disease). These scans will be taken after Courses 2 and 4 , then after every 3 courses until the therapy is finished, and once more at the end of therapy. Patients who show no signs of the disease will be given a total of up to 6 courses. Patients who have the disease may continue treatment until the disease gets worse. You will be taken off study if the disease gets worse or intolerable side effects occur. If you are removed from the study, you will be asked to have a follow-up CT scan or MRI and chest x-ray to evaluate the tumor.

THIS IS AN INVESTIGATIONAL STUDY. Paclitaxel is commercially available and approved for use in the treatment of ovarian cancer. Gleevec® is also commercially available and approved for use in the treatment of certain types of adult leukemias and stomach cancers. The combination of paclitaxel and imatinib mesylate is still investigational and has been approved for use in research only.

At least 51 and as many as 65 participants will take part in this study. All participants will be enrolled and treated at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed newly diagnosed (stage IIIC or IV) or recurrent (any stage) uterine papillary serous carcinoma. Patients with recurrent disease may not have been treated with taxanes in the past.
2. Patients may not receive concurrent radiotherapy while participating in this protocol.
3. Patients may have measurable or non-measurable disease.
4. Patients may have mixed endometrioid or clear cell components in addition to the serous histology.
5. Patients' tumor tissue must express one or more of the following biomarkers: c-Kit, PDGFR-B, or Abl. Positivity will be defined as 2+/3+ intensity in at least 10% of the tumor.
6. Patients must have pretreatment granulocyte count (i.e. segmented neutrophils and bands) of >/= 1,500/Fl, a hemoglobin level of >/= 9.0 gm/dl, and a platelet count of >/= 100,000/Fl.
7. Patients must have an adequate renal function as documented by serum creatinine of </=2.0 mg/dl.
8. Patients must have adequate hepatic function as documented by a serum bilirubin </=1.5mg/dl, regardless of whether patients have liver involvement secondary to tumor. Alanine aminotransferase (SGPT) and aspartate aminotransferase (SGOT) must be </=2.5x institutional upper limit of normal unless the liver is involved with tumor, in which case levels must be </=5x institutional upper limit of normal.
9. Zubrod performance status of 0, 1, or 2.
10. Patients should not have received prior chemotherapy or radiation (except palliative radiation) within the last 30 days.
11. Patients must have signed informed consent indicating that they are aware of the investigational nature of this study.

Exclusion Criteria:

1. Patients who have previously received imatinib mesylate or taxanes.
2. Patients with any active or uncontrolled systemic infection, including known HIV infection.
3. Patients with psychiatric disorders that would interfere with consent or follow-up.
4. Patients with New York Heart Association (NYHA) Class III/IV congestive heart failure, unstable angina or a history of myocardial infarction within the previous 6 months.
5. Patients with a history of prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least three years.
6. Oxygen-dependent lung disease.
7. Patients in whom corticosteroids are contraindicated.
8. Uncontrolled severe hypertension or uncontrolled diabetes mellitus.
9. Presence of clinically apparent central nervous system metastases or carcinomatous meningitis.
10. Patients with any form of chronic liver disease.
11. Patients with a history of seizures are ineligible. Patients receiving phenytoin, phenobarbital, or other anti-epileptic prophylaxis are ineligible.
12. Patients with any other severe concurrent disease, which in the judgment of the investigator, would make the patient inappropriate for entry into this study, including significant hepatic, renal, or gastrointestinal diseases.
13. Patients with a deep venous or arterial thrombosis (including pulmonary embolism) within 6 weeks of study entry.
14. Patients who are receiving therapeutic doses of warfarin or any blood thinning agent.
15. Patients with a history of non-compliance with medical regimens or who are considered potentially unreliable.
16. Pregnant or lactating women. Women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2003-12-29 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: December 29, 2003 to October 27, 2009. Recruitment was done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: The study was terminated early due to poor enrollment .
Groups:
- Phase I: Imatinib Mesylate 400 mg: Cohort One = Paclitaxel (Taxol) 175 mg/m^2 intravenous (IV) every 21 days + Imatinib Mesylate (Gleevec). Phase I Maximum Tolerated Dose (MTD) to be determined from escalating doses in subsequent cohorts: 400 (this arm, Cohort One), 500 (Cohort Two) or 600 mg (Cohort Three) orally daily.
- Phase I: Imatinib Mesylate 500 mg: Cohort Two = Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate 500 mg orally daily
- Phase I: Imatinib Mesylate 600 mg: Cohort Three = Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate 600 mg orally daily
- Phase II: Imatinib Mesylate MTD 500 mg: Phase II, Cohort 4 = Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate at MTD 500 mg orally daily
Period: Overall Study
Arm/Group | Phase I: Imatinib Mesylate 400 mg | Phase I: Imatinib Mesylate 500 mg | Phase I: Imatinib Mesylate 600 mg | Phase II: Imatinib Mesylate MTD 500 mg
Started | 4 | 6 | 2 | 5
Completed | 3 | 5 | 0 | 4
Not Completed | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Paclitaxel + Imatinib Mesylate: Phase I = Paclitaxel (Taxol) 175 mg/m^2 intravenous (IV) every 21 days + Imatinib Mesylate (Gleevec) 400, 500 or 600 mg orally daily
- Phase II: Paclitaxel + Imatinib Mesylate MTD 500 mg: Phase II = Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate at MTD 500 mg orally daily
- Total: Total of all reporting groups
Arm/Group | Phase I: Paclitaxel + Imatinib Mesylate | Phase II: Paclitaxel + Imatinib Mesylate MTD 500 mg | Total
Number analyzed (Participants) | 12 | 5 | 17
Age, Continuous [Median (Full Range); unit: years] | 62 [48 to 80] | 70 [60 to 77] | 64 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 11 | 4 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 10 | 4 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: Maximum Tolerated Dose (MTD) of Oral Imatinib Mesylate in Combination with Fixed Dose Paclitaxel where MTD of Imatinib Mesylate (mg/m^2 daily) to be determined with conventional 3+3 design, MTD is highest dose level in which 6 participants treated with at most 2 experiencing dose limiting toxicity (DLT). Study utilizes Common Terminology for Adverse Events Criteria (CTCAE) version 3.0 for adverse event reporting.
  Following cohorts of 3 at lower dose levels until 1 of 3 patients experiences DLT; if 1 of 3 patients experiences DLT at dose level, enter 3 additional patients at dose level, if only 1 of 6 patients experiences DLT at dose level, proceed to next higher dose level with cohort of 3; If 2 of 3 or 3 of 6 patients experience DLT, MTD has exceeded. Once DLT exceeded, treat another 3 patients at previous dose if there were only 3 patients treated at that dose level. MTD is highest dose level in which treated 6 patients with at most 2 experiencing the DLT.
Time Frame: Evaluated at 3 weeks (one cycle)
Population: One participant of 12 registered withdrew prior to receiving treatment.
Measure: Number; unit: participants
Groups:
- Imatinib Mesylate 400 mg: Cohort One = Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate 400 mg orally daily
- Imatinib Mesylate 500 mg: Cohort Two = Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate 500 mg orally daily
- Imatinib Mesylate 600 mg: Cohort Three = Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate 600 mg orally daily
Arm/Group | Imatinib Mesylate 400 mg | Imatinib Mesylate 500 mg | Imatinib Mesylate 600 mg
Number analyzed (Participants) | 4 | 6 | 2
participants | 0 | 1 | 2

2. Secondary Outcome: Number of Participants With Complete Response
Description: Complete Response (CR): Disappearance lesions, no evidence new lesions documented by 2 disease assessments> 4 weeks apart. Partial Response (PR):>30% decrease in sum longest dimensions (LD) all target measurable lesions reference baseline sum of LD; No progression non-target lesions & no new lesions; Documentation by 2 disease assessments >4 weeks apart; Progressive Disease (PD) (ANY of following): >20% increase in sum LD of target lesions reference smallest sum LD or appearance of new lesions within 8 weeks of study entry; Unequivocal progression on existing non-target lesions, other than pleural effusions without cytological proof of neoplastic origin, within 8 weeks of study entry also considered increasing disease. Death due to disease without prior objective documentation of progression; Global deterioration in health attributable to disease requiring change in therapy without objective evidence of progression. Stable disease: Any condition not meeting above criteria.
Time Frame: 6 weeks to 18 weeks; Best response achieved since study entry where measurable disease defined as => 1 lesion accurately measured in at least 1 dimension (longest dimension to be recorded)
Measure: Number; unit: participants
Groups:
- Participants With Measurable Disease; Participants With Non-Measurable Disease: Paclitaxel (Taxol) 175 mg/m^2 intravenous (IV) every 21 days + Imatinib Mesylate (Gleevec) 400, 500 or 600 mg orally daily or Phase II MTD 500 mg
Arm/Group | Participants With Measurable Disease | Participants With Non-Measurable Disease
Number analyzed (Participants) | 8 | 8
participants | 1 | 7

3. Secondary Outcome: Time to Tumor Progression
Description: Efficacy of Gleevec and Taxol in Participants defined by tumor progression for participants with measurable disease or recurrent non-measurable disease. Time to tumor progression defined as the time from date of initial treatment to first objective documentation of disease progression. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). After two cycles (6 weeks), participants will undergo clinical and radiographic (participants with measurable disease) tumor restaging or confirmation recurrent non-measurable disease. Evaluation of tumor response (for participants who already have the disease) determined by CT scan or MRI and chest x-ray (participants with chest disease).
Time Frame: Evaluation at at 6 weeks, tumor restaging continued up to 6 cycles (18 weeks) or until disease progression, whichever comes first
Population: Due to poor enrollment, the study was terminated early and no data collected for the Time to tumor progression outcome measure.
Arm/Group | Participants With Measurable Disease | Participants With Non-Measurable Disease
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Event collection with each 3 week cycle, up to 6 cycles (18 weeks).
Groups:
- Phase I: Imatinib Mesylate 400mg: Cohort One = Paclitaxel (Taxol) 175 mg/m^2 intravenous (IV) every 21 days + Imatinib Mesylate (Gleevec). Phase I Maximum Tolerated Dose (MTD) to be determined from escalating doses in subsequent cohorts: 400 (this arm, Cohort One), 500 (Cohort Two) or 600 mg (Cohort Three) orally daily.
- Phase II: Imatinib Mesylate 500 mg: Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate 500 mg orally daily
- Phase 1: Imatinib Mesylate 600 mg: Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate 600 mg orally daily
- Phase II: Imatinib Mesylate MTD 500 mg: Paclitaxel 175 mg/m^2 IV every 21 days + Imatinib Mesylate at MTD 500 mg orally
Arm/Group | Phase I: Imatinib Mesylate 400mg | Phase II: Imatinib Mesylate 500 mg | Phase 1: Imatinib Mesylate 600 mg | Phase II: Imatinib Mesylate MTD 500 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 2/2 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Imatinib Mesylate 400mg (N=4) | Phase II: Imatinib Mesylate 500 mg (N=6) | Phase 1: Imatinib Mesylate 600 mg (N=2) | Phase II: Imatinib Mesylate MTD 500 mg (N=5)
Fever w/o Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Fatigue (General disorders) | 4 | 6 | 2 | 3
Neuropathy (Nervous system disorders) | 3 | 3 | 2 | 3
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Pain - back (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 2 | 0 | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Neutrophils (Blood and lymphatic system disorders) | 4 | 6 | 1 | 4
Hemoglobin (Blood and lymphatic system disorders) | 2 | 6 | 1 | 4
Platelets (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 6 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 5 | 2 | 3
Vomiting (Gastrointestinal disorders) | 4 | 4 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Pain - abdomen (Gastrointestinal disorders) | 1 | 1 | 1 | 1
Pain - bone (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Rash - desquamation (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Mood alteration - anxiety (Nervous system disorders) | 1 | 1 | 0 | 0
Tinnitus (Eye disorders) | 1 | 0 | 0 | 0
Edema - facial (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Pain - pleura (General disorders) | 1 | 1 | 1 | 0
Heartburn (Gastrointestinal disorders) | 0 | 0 | 0 | 1
SGOT - elevated (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
SGPT - elevated (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes